CLINICAL TRIAL: NCT06658275
Title: Comparison of Constraint-Induced Movement Therapy And Bimanual Intensive Therapy Through Tele-rehabilitation For Upper Limb Functions In Children With Hemiplegic Cerebral Palsy
Brief Title: Comparison of Constraint-Induced Movement Therapy And Bimanual Intensive Therapy Through Tele-rehabilitation For CP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0234
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; neurological disorder; physiotherapy techniques; movement disorder; muscle spasticity
MeSH Terms: conditions — Cerebral Palsy; Nervous System Diseases; Movement Disorders; Muscle Spasticity | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Constraint-Induced Movement Therapy) (Experimental): Participants will undergo Constraint-Induced Movement Therapy(one hour), which will be administered by their parents under the guidance of a therapist through tele- rehabilitation for 3 days in a week for 8 weeks
  Interventions: Other: Constraint-induced movement therapy
- GROUP B (Bi-manual intensive therapy) (Experimental): Participants will undergo Bimanual therapy(one hour), which will be administered by their parents under the guidance of a therapist through tele-rehabilitation for 3 days in a week for 8 weeks.
  Interventions: Other: Hand Arm Bimanual Intensive Training -HABIT

INTERVENTIONS:
Other: Constraint-induced movement therapy — During the first routine checkup, therapists will educate caregivers on how to perform the exercises and activities at home. Caregivers will place the childrens less-affected hands in slings and guide them through exercises designed to engage their weaker, paretic hands. The sling will be fastened around the childrens trunks, with the end securely closed.After the initial session, the intervention will be provided by the caregiver at home, with progress monitored by the therapist through Zoom meetings or WhatsApp video calls. Children will engage in play-based activities as part of the CIMT program to improve upper limb functions.These activities will include painting, pin the tail on the donkey for sensory awareness and proprioception, card games, bubble activities, squeezing sponges, building towers with blocks, playing a curtained box game, using tongs, and picking up coins. Exercises will be gradually progressed from easier to more challenging tasks as the child improves.
  Arms: GROUP A (Constraint-Induced Movement Therapy)
Other: Hand Arm Bimanual Intensive Training -HABIT — For the Bimanual Intensive Training group, a strategy similar to HABIT will be used. At the first routine checkup, therapists will educate caregivers on the exercises, which will then be conducted at home. Caregivers will guide children through specially designed bimanual activities without slings, focusing on tasks like reaching, grasping, manipulation, releasing, and bearing weight on the upper limb. Progress will be monitored remotely through Zoom or WhatsApp video calls.Exercises will include catching and throwing a ball to improve reaching, grasp, and release; squeezing a textured ball for sensory awareness and sustained grip; stabilising and reorienting paper while drawing and cutting to enhance forearm supination and wrist extension. Additional tasks like sticker peeling for pincer grip and dough playing for hand manipulation will also be included.Exercises will progress from easy to more difficult as the child improves
  Arms: GROUP B (Bi-manual intensive therapy)

SUMMARY:
Cerebral palsy is a neurological condition affecting movement and posture, caused by non-progressive brain disruptions occurring during fetal development. Constraint-induced movement therapy (CIMT) significantly improves arm and hand function in children with hemiparetic cerebral palsy by using intensive therapy sessions and restricting the unaffected limb to develop new motor skills. Bimanual therapy involves using both hands repeatedly to perform functional tasks, rather than relying on just one hand. Tele-rehabilitation (TR) is an affordable method of providing remote rehabilitation services through telecommunication technologies like smartphones and media applications. The aim of the study is to compare the effectiveness of CIMT and bimanual therapy delivered via tele-rehabilitation for improving upper limb function in children with cerebral palsy.

This randomized clinical trial will be conducted at Mubarik Medical Complex, Sargodha, Pakistan, with a sample size of 65. Participants will be randomly allocated into two groups using an online randomization tool, Group A will receive constraint-induced movement therapy (CIMT) intervention for 60 minutes, and Group B will receive bimanual therapy intervention for 60 minutes. Each participant will undergo treatment for three days a week on alternate days for eight weeks.

Spasticity will be assessed by using the Modified Ashworth Scale. The Quality of Upper Extremity Skills Test (QUEST) will evaluate dissociated movement, grasp, protective extension, and weight bearing, while the Tele-Rehabilitation Satisfaction Survey (TeSS) is designed to evaluate the experiences and satisfaction levels of patients or caregivers who have participated in tele-rehabilitation programs. Measurements will be taken at baseline, 4th week, 8th week, and at 12th week after discontinuation of treatment. The data will be entered and assessed using SPSS 26. For between-group analysis of parametric data, the independent t-test will be used, while non-parametric data will be analyzed using the Mann-Whitney test. Within-group comparisons will be conducted using repeated measures ANOVA for parametric data and Friedman ANOVA for non-parametric data.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-12 years.
* Children with hemiplegic cerebral palsy with mild to moderate hand involvement.
* Ability to extend wrist >20° and fingers at the metacarpophalangeal joints

  >10° from full flexion
* Demonstrated ability to follow instructions during screening and complete the testing.
* Spasticity does not exceed a score of 1 or 1+ on the Modified Ashworth Scale

Exclusion Criteria:

* Health problems unassociated with CP.
* Visual problems interfering with treatment.
* Active or unstable seizures.
* Orthopedic surgery on the more affected hand within the last year.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Quality Of Upper Extremity Skills Test (QUEST) | 8 weeks
  The Quality of Upper Extremity Skills Test (QUEST) was developed in 1991 specifically to address the needs of children with spastic cerebral palsy. It is a criterion-referenced assessment tool designed to measure the quality of upper limb movements. The test comprises 34 items, which are organized into four distinct domains. These domains collectively evaluate various aspects of upper extremity function. Administering and scoring the QUEST typically takes between 30 and 45 minutes.
Telehealth Satisfaction Scale | 8 weeks
  The Telehealth Satisfaction Scale (TeSS) is a standardized tool designed to assess patient satisfaction with telehealth services. It evaluates aspects such as the quality of care, ease of use of telehealth technology, interaction with healthcare providers, and overall telehealth experience.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, PhD-PT, Study Chair — Riphah International University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gorter JW, Rosenbaum PL, Hanna SE, Palisano RJ, Bartlett DJ, Russell DJ, Walter SD, Raina P, Galuppi BE, Wood E. Limb distribution, motor impairment, and functional classification of cerebral palsy. Dev Med Child Neurol. 2004 Jul;46(7):461-7. doi: 10.1017/s0012162204000763. PMID 15230459